CLINICAL TRIAL: NCT04145232
Title: Development of AImmune Technology as a Bioinformatic Component of Diagnostic Tests Used in Cancer Immunotherapy
Brief Title: AImmune - Artificial Intelligence Algorithm for Identification of Immunogenic Neoepitopes of Cancer to Predict and Boost Patient's Response to Immunotherapies.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ardigen (Industry)
Collaborators: Małopolskie Centre of Entrepreneurship (Unknown)
Responsible Party: Sponsor
Other Study IDs: A.I.mmune; RPMP.01.02.01-12-0301/17 (Other Grant/Funding Number: Małopolskie Centre of Entrepreneurship)
Record Dates: First submitted 2019-10-29; First posted 2019-10-30 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-08

CONDITIONS: Non Small Cell Lung Cancer; Neoepitopes; Neoantigens; Immunotherapy; Next Generation Sequencing (NGS); Personalized Neoantigen Cancer Vaccine
Keywords: Cancer; Non Small Cell Lung Cancer; Neoepitopes; Neoantigens; Immunotherapy; Nivolumab; Ipilimumab; Atezolizumab; Neoantigen cancer vaccine; Personalized neoantigen cancer vaccine; FFPE; PBMC; Stool; Immuno-Oncology; Next generation sequencing (NGS)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms | interventions — Blood Specimen Collection; Nivolumab; Ipilimumab; atezolizumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — biopsy (FFPE), peripheral blood samples (PBMC) and stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NSCLC: This cohort will consist of 30 patients with non-small cell lung cancer (NSCLC).
  Interventions: Biological: Collection of biopsy (FFPE), blood (PBMC) and stool

INTERVENTIONS:
Biological: Collection of biopsy (FFPE), blood (PBMC) and stool — Patients receiving routine treatment (immunotherapy using anti-PD1 / anti-PDL1 and / or anti CTLA4 antibodies), financed by the Polish National Health Fund (NFZ).
  Other Names: Nivolumab; Ipilimumab; Atezolizumab

SUMMARY:
The goal of the project is to develop and validate A.I.mmune technology. It performs complex analyses of patients' tumor and immune system state using data derived from next-generation sequencing of tumor and healthy tissue to identify cancer neoantigens, which are likely to elicit an immune response.

A key challenge to be solved using the technology is to predict for each patient which neoepitopes are not only likely to bind to HLA or be presented on the tumor cell surface, but also will be recognized by the T-cell receptor and create the immunogenic response. The presence of such epitopes is required for immunotherapy by immune checkpoint inhibition to have an effect on the disease. Knowledge of those epitopes enables therapeutic strategies to boost the immune response by designing personalized cancer vaccines and adoptive cell therapies.

The samples and data collected in this clinical study will be used for clinical validation of A.I.mmune technology. For all patients treated with immunotherapy (using anti-PD1 / anti-PDL1 and / or anti-CTLA-4 antibodies) peripheral blood samples (PBMC) and biopsy (FFPE) collection will be performed before treatment. Samples will be sequenced by next-generation sequencing platform. In parallel, the investigators will also collect samples of stool (one sample before the start of immunotherapy) and follow-up information of responses to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Men or women ≥18 years of age.
* Patients with non-small cell lung cancer.
* Patients with informed consent to participate in the study.
* Patients receiving routine treatment (immunotherapy using anti-PD1 / anti-PDL1 and / or anti CTLA4 antibodies), financed by the Polish National Health Fund (NFZ).
* The applied immunotherapy should be the first or second line of treatment.

Exclusion Criteria:

* Patients who are unable to understand, read and / or sign informed consent.
* Patients who can not collect stools.
* Patients with fecal transplant.
* The applied immunotherapy is not the first or second line of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving routine treatment.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-06-13 (Actual); Primary Completion 2020-10-15 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
Number of Responders and Non-responders on immunotherapy (evaluated using RECIST 1.1 criteria) | Up to 6 months
  Standard follow-up care after cancer treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Stepniak, Principal Investigator — Ardigen
Locations (1):
- University Clinical Centre in Gdansk, Gdansk, Poland